CLINICAL TRIAL: NCT00626912
Title: PRET: Patients Prone to Recurrence After Endovascular Treatment. A Randomized Trial Comparing Platinum and Hydrogel-coated Coils
Brief Title: PRET: Patients Prone to Recurrence After Endovascular Treatment
Acronym: PRET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ND07.001
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2016-07

CONDITIONS: Intracranial Aneurysm; Subarachnoid Hemorrhage
Keywords: large aneurysm; recurrence; hydrocoil
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): platinum coils
  Interventions: Procedure: endovascular coil embolization
- 2 (Active Comparator): hydrogel coils
  Interventions: Procedure: endovascular coil embolization

INTERVENTIONS:
Procedure: endovascular coil embolization — standard endovascular coil embolization with or without adjunct techniques
  Other Names: platinum coil; hydrogel coil

SUMMARY:
The PRET study aims at comparing two types of coils used in the endovascular treatment of intracranial aneurysms. The first type made of platinum has been used for more than 15 years. The other, referred to as hydrocoil, containing in addition to platinum a polymer layer that expands when in contact with blood, has been in use since 2002. The hypothesis of the PRET study is that the newer hydrocoil will be more effective and yet as safe as the older platinum coil.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting at least one aneurysm 'prone to recurrence after endovascular treatment' (PRET), defined for the sake of this study as:

  * PRET-1: One ruptured or unruptured aneurysm, never treated, with a dimension ≥10mm (longest axis, including thrombosed portions of large or giant aneurysms); for ruptured lesions, patients should be in WFNS grade I, II or III.
  * PRET-2: an Aneurysm presenting a major recurrence after previous coiling; and judged by the neurovascular team to require elective treatment.
* The anatomy of the lesion is such that endovascular treatment is possible with both types of coils (not necessarily certain or probable)
* The endovascular physician is content to use either type of coils (platinum or hydrogel-coated coils) but no other type of coils
* Patient is 18 or older
* Life expectancy is more than 2 years

Exclusion Criteria:

* Presence of other aneurysms requiring treatment during the same session
* Patients with associated cerebral arteriovenous malformations
* When parent vessel occlusion, without simultaneous endosaccular coiling of the aneurysm, is the primary intent of the procedure
* Any absolute contraindication to endovascular treatment, angiography, or anaesthesia such as severe allergies to contrast or medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2007-06; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean RAYMOND, MD, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); Daniel ROY, MD, Study Director — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (32):
- United States (18):
  - Shands - University of Florida Hospital, Gainesville, Florida
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississipi Health Care, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Washington University in St Louis, St Louis, Missouri
  - University of Buffalo (SUNY), Buffalo, New York
  - Stony Brook University Medical Center (SUNY), Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - The Methodist Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal - Notre Dame Hospital, Montreal, Quebec
- Instituto de Neurocirugía Dr. Asenjo, Santiago, Chile
- France (6):
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU Henri Mondor - Hôpital Henri Mondor, Créteil
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU Nancy-Hôpital Central, Nancy
  - CHU de Nantes - Hôpital Guillaume et René Laennec, Nantes
  - Centre Hospitalier Sainte Anne, Paris
- Kobe City Medical Center General Hospital, Kobe, Japan
- United Kingdom (3):
  - Leeds General Infirmary, Leeds
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Queens Medical Centre, Nottingham

REFERENCES:
- [Derived] Naggara O, Darsaut T, Trystram D, Tselikas L, Raymond J. Unruptured intracranial aneurysms: why we must not perpetuate the impasse for another 25 years. Lancet Neurol. 2014 Jun;13(6):537-8. doi: 10.1016/S1474-4422(14)70091-2. No abstract available. PMID 24849854

RESULTS

PARTICIPANT FLOW:
Groups:
- Platinum Coils: Endovascular coil embolization with standard platinum coils
- Hydrogel Coils: Endovascular Coil embolization with Hydrogel Coils
Period: Overall Study
Arm/Group | Platinum Coils | Hydrogel Coils
Started | 222 | 225
Completed | 220 | 215
Not Completed | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Platinum Coils: Endovascular coil embolization with standard platinum coils
  endovascular coil embolization: standard endovascular coil embolization with or without adjunct techniques
- Hydrogel Coils: Endovascular coil embolization with hydrogel coils
  endovascular coil embolization: standard endovascular coil embolization with or without adjunct techniques
- Total: Total of all reporting groups
Arm/Group | Platinum Coils | Hydrogel Coils | Total
Number analyzed (Participants) | 222 | 225 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 57 (11) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 165 | 319
  Male | 68 | 60 | 128
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 75 | 61 | 136
  United States | 112 | 126 | 238
  Japan | 3 | 1 | 4
  United Kingdom | 10 | 12 | 22
  France | 15 | 18 | 33
  Chile | 7 | 7 | 14
Ruptured aneurysms (Number) [Count of Participants; unit: Participants] | 39 | 40 | 79
Aneurysm size (mean (SD)) [Mean (Standard Deviation); unit: millimeters] | 11.3 (5.8) | 10.7 (5.3) | 11.0 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate of Target Aneurysm.
Description: 1. major angiographic recurrence of the lesion or the presence of a residual aneurysm at last angiographic follow-up, as determined by the core laboratory, blinded to treatment allocation;
  2. retreatment of the same aneurysm by endovascular or surgical means during the 18-month follow-up period;
  3. an intracranial bleeding episode, or the occurrence or progression of a mass effect in relation to the treated aneurysm during the follow-up period, as determined by the blinded Adverse Event Committee.
Time Frame: 18 months
Population: For the Platinum coils population (222):
  Primary outcome available for 220/222 (could not attribute primary outcome for 2 participants)
  For the Hydrogel coils population (225):
  Withdrawn by physician right after Registration: 3/225 (remaining 222) Primary outcome available for 215/222 (could not attribute primary outcome for 7 participants)
Measure: Count of Participants; unit: Participants
Groups:
- Platinum Coils: platinum coils
  endovascular coil embolization: standard endovascular coil embolization with or without adjunct techniques
- Hydrogel Coils: hydrogel coils
  endovascular coil embolization: standard endovascular coil embolization with or without adjunct techniques
Arm/Group | Platinum Coils | Hydrogel Coils
Number analyzed (Participants) | 220 | 215
Participants | 102 | 103

2. Secondary Outcome: Mortality Rate
Description: Number of participants dead - All causes
Time Frame: 18 months
Population: For the Platinum coils population (222):
  Secondary outcome measure applies to 222 participants.
  For the Hydrogel coils population (225):
  Withdrawn by physician right after Registration: 3/225 (remaining 222). Secondary outcome measure applies to 222 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum Coils | Hydrogel Coils
Number analyzed (Participants) | 222 | 222
Participants | 3 | 13

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants having experienced one or several Adverse Events. This measure is the number of participants having experienced Serious Adverse Events plus those having experienced other (not including Serious) Adverse Events.
Time Frame: 18 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum Coils | Hydrogel Coils
Number analyzed (Participants) | 222 | 222
Participants | 37 | 41

4. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants having experienced one or several Serious Adverse Events
Time Frame: 18 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum Coils | Hydrogel Coils
Number analyzed (Participants) | 222 | 222
Participants | 20 | 25

ADVERSE EVENTS:
Time Frame: 18 months
Description: an Adverse Event is defined as an event of any severity being possibly or probably related to the disease or the treatment and happening at any time during the 18-month follow-up period. The independent Adverse Event Committee was responsible for the attribution of Adverse Events.
Arm/Group | Platinum Coils | Hydrogel Coils
All-Cause Mortality (participants affected / at risk) | 3/222 | 13/222
Serious Adverse Events (participants affected / at risk) | 20/222 | 25/222
Other Adverse Events (participants affected / at risk) | 17/222 | 16/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum Coils (N=222) | Hydrogel Coils (N=222)
sub-arachnoid hemorrhage (Vascular disorders) | 2 (2) | 2 (2)
Mass Effect (Vascular disorders) | 1 (1) | 1 (1)
stroke (Vascular disorders) | 2 (2) | 2 (2)
subdural hematoma (Vascular disorders) | 0 (0) | 1 (1)
non neurologic (Vascular disorders) | 2 (2) | 0 (0)
Retreatment related (Surgical and medical procedures) | 0 (0) | 5 (5)
periprocedure event (Surgical and medical procedures) | 13 (13) | 14 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum Coils (N=222) | Hydrogel Coils (N=222)
Transient Ischemic Attack (Vascular disorders) | 0 (0) | 1 (1)
Mass Effect (Vascular disorders) | 1 (1) | 0 (0)
Inflammatory (Vascular disorders) | 2 (2) | 0 (0)
Non neurologic (Vascular disorders) | 1 (1) | 1 (1)
Retreatment related (Surgical and medical procedures) | 3 (3) | 0 (0)
Periprocedure event (Surgical and medical procedures) | 10 (10) | 14 (14)

LIMITATIONS AND CAVEATS:
Operators could not be blinded to coil type. This may have affected case selection, coil selection, and completeness of the coiling procedure. Aneurysm volumes were not directly measured but extrapolated from aneurysm dimensions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No